CLINICAL TRIAL: NCT06769854
Title: Defining the Safety and Efficacy of POSterIor Tibial NeRve StimulatiON in Children
Acronym: POSITRON-C
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chi Dang Hornik (Other)
Collaborators: Duke Clinical Research Institute (Other); The Emmes Company, LLC (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Chi Dang Hornik, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114395; HHSN275201800003I (Other Grant/Funding Number: National Institute of Child Health and Human Development)
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome
Keywords: PTNS; Overactive Bladder; percutaneous tibial nerve stimulation; Urgent PC; urinary urgency; urinary incontinence; urinary frequency; OAB; urinary urge; Urinary Bladder; Urinary Bladder Diseases; Urologic Diseases; Pediatrics
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Urinary Bladder Diseases; Urologic Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single-arm cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-Arm Cohort (Experimental): Single Arm Cohort: (n=50) PTNS treatment weekly over 30 minutes for a total of 12 weekly sessions.
  Interventions: Device: Urgent PC

INTERVENTIONS:
Device: Urgent PC — PTNS is a technique of electrical neuromodulation used primarily for treating OAB. The procedure for PTNS consists of the insertion of a fine needle above the medial malleolus near the posterior tibial nerve followed by the application of low-voltage electrical stimulation that produces sensory and motor responses.
  Other Names: Non-drug, non-surgical treatment for overactive bladder; PRC 26348 - V1.00

SUMMARY:
The purpose of this study is to find out if overactive bladder (OAB) can be safely treated by stimulating a nerve near the ankle. This procedure is called percutaneous tibial nerve stimulation (PTNS). It will be done by a device called the Urgent PC. The Urgent PC works by sending weak electrical signals through a thin needle to the nerve near the ankle. Stimulating this nerve may change bladder control.

DETAILED DESCRIPTION:
This study is a single-arm, open label, prospective, multicenter study of 50 participants aged 5-21 years with OAB. Participants will undergo outpatient PTNS sessions per routine clinical care using Urgent PC once weekly for 12 weeks. Patients, parents and clinicians will not be blinded to treatment or assessments during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-21 years old (inclusive)
2. Obtained legally effective informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization from the participant or the participant's parent/legal guardian/legally authorized representative (LAR)
3. Minor participant is willing and able to provide assent (as applicable)
4. History of primary or secondary non-neurogenic OAB as defined by a VDES score of ≥11 and a positive modified bother score within 30 days of consent
5. Has previously tried and failed standard urotherapy and at least one anticholinergic or beta-3 adrenergic agonist
6. Adequate fluid intake for age as reported by participant or parent/legal guardian/LAR
7. Micturition frequency of at least 8 times (mean)/day for at least 4 weeks prior to enrollment
8. At least 1 daytime incontinence episode (mean)/day for at least 4 weeks prior to enrollment
9. If on allowed treatment for OAB, stable dose for at least 30 days prior to screening and willingness to continue that dose for the duration of the study

Exclusion Criteria:

1. Known or apparent untreated anatomical abnormality of the lower urinary tract (e.g., untreated ureterocele)
2. Known neurogenic bladder (e.g., spina bifida, history of spinal cord injury, tethered cord)
3. Presence of local skin lesions (e.g., rash, skin infections) on the medial surfaces of both ankles at the time of consent
4. Metal implants in the medial ankle area
5. Pacemakers or implantable defibrillators
6. History of excessive bleeding
7. Nerve damage that may impact the percutaneous tibial nerve or pelvic floor function
8. History of chemodenervation of the bladder (e.g., via intravesical instillation or intradetrusor injection of botulinum toxin)
9. Known current, untreated UTI
10. Current or previous pregnancy at screening or planned pregnancy during the duration of the study, for females of childbearing potential
11. Any condition that, in the judgment of the investigator or treating clinician, precludes participation because it could affect participant safety
12. Previous treatment with this device or participation in this study or in any other study for the treatment of OAB
13. High-grade vesicoureteral reflux (grades 4-5)
14. Diagnosed diabetes insipidus (pituitary, nephrogenic, or acquired)
15. Stage 4-5 chronic kidney disease (CKD) (since device may further disrupt or exacerbate abnormal urine flow)
16. Significant post-void residual defined as >60 mL
17. Initiation of or change of OAB treatment during screening or the duration of the study.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2027-04-01 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
The frequency of select safety Events of Special Interest. | Weekly, Week 1 through Week 16
  1. Electrode site reaction (bruising, bleeding, hematoma, or persistent erythema at the electrode site)
  2. Electrode site infection
  3. Repeated post-void residual >60 mL (at ≥ 2 consecutive visits)
  4. Urinary tract infection
  5. Urinary retention/obstruction
  6. Toe numbness
  7. Stomach and leg cramps
Change in maximum voided volume on the Bladder Diary | Week 1, Week 12
  The Bladder Diary is a paper diary recommended by the International Children's Continence Society that will be completed by the parent/guardian/LAR or participant. The Bladder Diary includes the following variables: fluid intake, number of voids, volume of voids, degree of urgency, number of incontinent episodes.

SECONDARY OUTCOMES:
Proportion of children who experienced complete response, no response, or partial response on the Vancouver Dysfunctional Elimination Survey (VDES) | Screening, Weekly (Week 1 through Week 12)
  The VDES is a validated questionnaire that was developed for diagnosing dysfunctional elimination syndrome. The survey uses a five-point Likert scale to score symptoms of bladder dysfunction. Each question is scored on a scale of 0-4, with 0 indicating no complaints and 4 indicating severe symptoms. The total score ranges from 0-52, with higher scores indicating more severe symptoms. The question about voiding frequency is scored differently from the other questions. A neutral choice of five to six urination per day is scored as 0. A urinary frequency of one to two times or more than eight times a day is scored as 4. A urinary frequency of three or four and seven or eight times a day is scored as 2. A cutoff score of 11 is used for patients and 9 for parents to diagnose dysfunctional voiding. The VDES is completed by the parent/legal guardian if participants are < 9 years old and by participants if they are ≥ 9 years old.
Change in OAB symptoms (Urgency, Frequency and Daytime Incontinence) reported on the VDES | Screening, Weekly (Week 1 through Week 12), Week 16, Week 36
  Change in OAB symptoms will be evaluated from the symptom questions on the VDES survey assessing Urgency, Frequency and Daytime Incontinence. The survey uses a five-point Likert scale to score symptoms of bladder dysfunction. Each question is scored on a scale of 0-4, with 0 indicating no complaints and 4 indicating severe symptoms. The total score ranges from 0-52, with higher scores indicating more severe symptoms. The question about voiding frequency is scored differently from the other questions. A neutral choice of five to six urination per day is scored as 0. A urinary frequency of one to two times or more than eight times a day is scored as 4. A urinary frequency of three or four and seven or eight times a day is scored as 2. A cutoff score of 11 is used for patients and 9 for parents to diagnose dysfunctional voiding. The VDES is completed by the parent/legal guardian if participants are < 9 years old and by participants if they are ≥ 9 years old.
Proportion of children who develop a febrile UTI | Weekly, Week 1 through Week 12
  Febrile UTI occurrence, defined as:
  • Fever > 101.5°F (> 38.6°C); and >50,000 colony forming units (CFU)/mL of 1 or more speciated organisms; and 10 white blood cells per higher power field (WBC/HPF) on urine microscopy and/or leucocyte esterase > 2+ on dipstick; and At least 1 of the following symptoms: Gross hematuria (defined as pink or red urine, not a spot of blood on a catheter) OR Abdominal, suprapubic, or flank pain or tenderness OR New or worsening incontinence OR New or worsening urinary urgency, frequency, or hesitancy OR Nausea/vomiting OR Pain with urination OR Malodorous/cloudy urine.
The change of Pediatric Incontinence Quality of Life (PINQ) score | Week 1, Week 6, Week 12, Week 16, and Week 36
  The Pediatric Incontinence Quality of Life (PINQ) is a 20-item, self-reported questionnaire that evaluates the QoL of children who have urinary incontinence. Each item is scored on a 5-point Likert scale, with 1 being "no" and 5 being "always". The total score ranges from 20 to 100 points. A higher score indicates a better QoL that is less affected by urinary symptoms. The PINQ is validated for use in children 6-17 years old and has been used in studies of participants up to 30 years old.21,25 The PINQ will be completed by the parent/legal guardian/LAR if participants are < 9 years old and by participants if they are ≥ 9 years old.
The percent of study visits attended within the protocol specified window from baseline through Week 12 | Screening, Weekly (week 1 through week 12)
  The percent of study visits attended within the protocol specified window from baseline through Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hornik, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: Yes
All data collected is uploaded into the National Institute of Health Data Repository (DASH) at the end of the study (de-identified).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be uploaded to the repository within 2 years of study completion. It will be maintained in the repository indefinitely.
Access Criteria: In order to have access, researchers have to complete a Data access request. NICHD will review the request and either approve or deny it. IRB approval must be obtained by the researcher to access the data. https://dash.nichd.nih.gov/Resource/DataRequestChecklist
URL: https://dash.nichd.nih.gov/